CLINICAL TRIAL: NCT06189846
Title: Prospective Study Incorporating LUMENEYE Rectoscope for Assessment on Tumor Response After Total Neoadjuvant Treatment in Rectal Cancer
Brief Title: Lumeneye Rectoscope for Assessment on Tumor Response After Total Neoadjuvant Treatment in Rectal Cancer
Acronym: LUMEVAL
Status: Recruiting | Type: Observational
Sponsor: Bordeaux Colorectal Institute Academy (Other)
Responsible Party: Sponsor
Other Study IDs: BCIA 2023/02
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: International Cohort — Assessing tumour response following neoadjuvant treatment in rectal cancer include :
  * Digital rectal examination
  * Rectal MRI
  * Rectoscopy ( Lumeneye device)
  The monitoring of tumour response intervals up to 6 months following completion of the neoadjuvant treatment at 8 weeks, at 16 weeks, at 24 weeks after the end of neoadjuvant treatment.

SUMMARY:
The objective of this prospective international cohort is to evaluate the LUMENEYE rectoscope for assessment on tumor response after total neoadjuvant treatment in rectal cancer.

Patients included in this study will be patients who initially will be good candidates for organ preservation. The participating centers are all expert centers in tumor assessment.

All patient assessments after neoadjuvant treatment for rectal adenocarcinoma will be included in each centre.

DETAILED DESCRIPTION:
The recent validation of the Total Neoadjuvant Treatment (TNT) protocol and the improvement of techniques for evaluating tumor response are two major factors in the development of organ preservation in rectal cancer.

Although recent publications have shown promising results of the two organ preservation strategies, Watch & Wait and Local excision, with a low oncological risk, some challenges remain to be addressed before the generalization of rectal preservation in clinical practice.

Among these challenges, the improvement of patient selection and methods for evaluating tumor response appear necessary. The monitoring scheme for the tumor response has not yet been clearly established, but a 6 months programme of tumor response assessment has been recently published (Boubaddi EJSO 2023). Monitoring must consist of a clinical assessment (rectal examination and/or rectoscopy) and additional morphological examinations (rectal MRI) every two months.

Tumor response after neoadjuvant treatment by MRI (TRG 1-5, Tumor Regression Grade) is established as a reliable method of tumor response assessment and accurate diagnosis of complete clinical response. However, discrepancies between clinical examination and radiological MRI may exist and patients undergoing watch-and-wait who develop local regrowth due to mistake in initial tumour response assessment are at higher risk for development of distant metastases (Sao Juliao DCR 2023) with a poor impact on long term oncological results.

The development of the LumenEye digital rectoscope by the SurgEase company enables a comfortable and efficient scoping for the user and the patient (Lewis J BJGP Open 2022). With high quality images of Full HD images and video associated with a secure and connected intuitive software platform, this endoscope can have its place in the monitoring of tumor response.

The contribution of this technology to the monitoring of the tumor response needs to be assessed. This medical device is CE marked and used in its intended purpose.

The objective of this study is to evaluate the complete and/or nearly complete response with LumenEye digital rectoscope.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Histologically confirmed diagnosis of adenocarcinoma of the rectum,
* Patient who received radiotherapy and chemotherapy (TNT) or immunotherapy
* Stage cT2T3
* cN0 or cN1 (≤ 3 positive LN or size ≤ 8 mm)
* no metastases
* Baseline Tumour size ≤ 5 cm (MRI)
* Baseline Tumour ≤ 8 from anal verge
* Ability to consent.
* Oral agreement after reading information letter

Exclusion Criteria:

* Tumour cT1 or cT4
* Baseline Tumour size > 5cm
* Invaded external sphincter or levator muscle
* Tumour cN2 (> 3 positive LN or size > 8 mm)
* Metastasis
* History of Inflammatory bowel disease
* Patient with a history of pelvic radiotherapy or chemotherapy
* Pregnant patients
* Protected adults (individuals under guardianship by court order).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These are patients with small rectal cancer, initially good candidates for organ preservation and whose evaluation is done by clinical and radiological examination and with the Lumeneye rectoscope
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The rate of complete and/or nearly complete response | From 8 weeks to 24 weeks after the end of radiotherapy
  To evaluate the complete and/or nearly complete response with LumenEye digital endoscopescope

SECONDARY OUTCOMES:
Agreement for grading rectal tumour response between the endoscopic and MRI assessment of tumour response | From 8 weeks to 24 weeks after the end of radiotherapy
  To evaluate the concordance between the endoscopic and MRI assessment of tumor response
Agreement for grading rectal tumour response between the clinical and endoscopic assessment of tumour response | From 8 weeks to 24 weeks after the end of radiotherapy
  - To evaluate the concordance between the clinical and endoscopic assessment of tumor response.
Agreement for grading rectal tumour response between the clinical and MRI assessment of tumour response. | From 8 weeks to 24 weeks after the end of radiotherapy
  To evaluate the concordance between the clinical and MRI assessment of tumor response.
Interobserver agreement for grading rectal tumour response using a digital rectoscope platform | From 8 weeks to 24 weeks after the end of radiotherapy
  To assess the interobserver reproducibility of endoscopic response with LumenEye digital endoscope within 6 months after the end of neoadjuvant treatment.
Rate of changing attitude after using the digital rectoscope platform (intra-observer changing management). | From 8 weeks to 24 weeks after the end of radiotherapy
  To evaluate the contribution of the digital ectoscope platform in the surgeon's decision-making

CONTACTS AND LOCATIONS:
Overall Officials: Quentin DENOST, Study Director — Bordeaux Colorectal Institute
Locations (8):
- France (4):
  - Clinique Tivoli-Ducos - Bordeaux Colorectal Institute, Bordeaux
  - Hôpital Européen de Marseille, Marseille
  - Hôpital Saint-Antoine - APHP, Paris
  - CHU de ROUEN, Rouen
- Humanitas Research Hospital, Milan, Italy
- Amsterdam UMC, Amsterdam, Netherlands
- University Hospital Vall D'Hebron, Barcelona, Spain
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No